CLINICAL TRIAL: NCT06269809
Title: Temporary Artery Clipping for Robotically-assisted Myomectomy, a Multicentric Randomized Controlled Trial
Acronym: TACROM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Amsterdam UMC, location VUmc (Other); Bichat Hospital (Other); Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: s67279
Record Dates: First submitted 2023-07-13; First posted 2024-02-21 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Fibroid Uterus
Keywords: myomectomy; fibroid; myoma; blood loss; temporary artery clipping; hemostatic measures
MeSH Terms: conditions — Leiomyoma; Myoma; Hemorrhage

STUDY DESIGN:
Intervention Model Description: Multicentric non-blinded randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Temporary artery clipping (Experimental): Patients undergoing a robotically-assisted myomectomies, with temporary clipping of the uterine arteries and the utero-ovarian ligmants.
  Interventions: Procedure: Temporary clipping of the uterine arteries and the utero-ovarian ligmants.
- Control (Active Comparator): Patients undergoing a robotically-assisted myomectomies, without temporary clipping of the uterine arteries and the utero-ovarian ligmants.
  Interventions: Procedure: No temporary clipping of the uterine arteries and the utero-ovarian ligmants.

INTERVENTIONS:
Procedure: Temporary clipping of the uterine arteries and the utero-ovarian ligmants. — Temporary clipping of the uterine arteries and the utero-ovarian ligaments using laparoscopic clips/bulldog clamps, during robotically assisted myomectomy.
  Arms: Temporary artery clipping
Procedure: No temporary clipping of the uterine arteries and the utero-ovarian ligmants. — Robotically assisted myomectomy, for which no temporary clipping of the uterine arteries and the utero-ovarian ligaments
  Arms: Control

SUMMARY:
This study aims to investigate the efficacy of temporary clipping of the uterine artery and utero-ovarian ligament during robotically assisted myomectomy (RAM) for uterine fibroids. While RAM is increasingly used for myomectomy, bleeding control remains challenging. Temporary clipping of arteries has shown promise in conventional laparoscopy but has not been studied in RAM. This randomized controlled trial will assess primary endpoints such as estimated blood loss, need for transfusion, and hemoglobin drop, alongside secondary outcomes like complication rates and operation time.

DETAILED DESCRIPTION:
Uterine fibroids, also known as myomas or leiomyomas, are benign smooth muscle neoplasms of the uterus. Uterine fibroids are the most common neoplasms affecting women of reproductive age (up to 70-80% at the age of 50)(1). As fibroids grow, they may induce clinical problems such as menorrhagia, abdominal pain, or infertility.(2,3) Removal of uterine fibroids (myomectomy) is a gynaecological surgical procedure performed most frequently through laparotomy or minimally invasive surgery such as conventional laparoscopic or robotically assisted surgery. Because of the straight-stick instruments with limited degree of freedom, the excision and suturing of the myoma can be rather cumbersome, not in the least because myomectomies may be associated with relatively profuse peri-operative bloodloss. Owing to its enhanced 3D vision and wristed instruments, robotically assisted surgery may be a more suitable surgical technique, especially in the case of multiple myomas, large myomas or posterior localization. Consequently, in recent years a gradual shift has been seen to the use of robotically assisted myomectomies.

However, control of the bleeding during a myomectomy can be a challenge, even in the hands of an experienced robotic surgeon. Various strategies have been developed to combat this scenario; including rectal or IV misoprostol, intramyometrial injection of bupivacaine with epinephrine or vasopressin, , tranexaminic acid IV or various ligation strategies. There is moderate quality evidence for some of these interventions. Recently, the use of clips to temporary occlude the uterine artery for myomectomy with conventional laparoscopy for prevention of blood loss was validated in several studies, including 2 randomized controlled trials. To enhance hemostasis, recent articles described a technique to temporary clip both the uterine artery and infundibulopelvic artery with conventional laparoscopy, also resulting in fewer intra-operative bleeding compared to no artery clipping. The possible benefit of these ligation technique has never been studied in the setting of robotically-assisted myomectomies. On the one hand, RAM may involve more complex cases due to myoma size, localization or multiple myomas, and on the other hand, bleeding control may also be better with robotic surgery. This makes a prediction of the usefulness of this technique difficult, in terms of reducing blood loss.

Estimated blood loss remains a difficult outcome to reliably quantify, especially when using only visual parameters. During RAM, often only suction is used, making the estimation easier in comparison to open surgery, for which a variety of compresses and suction is used. This study will work with multiple primary endpoints, combining estimated blood loss over 500 mL, the need for a peri-operative blood transfusion or a hemoglobin drop exceeding 2 g/dL.

Other secondary outcomes will include complication rate, the operation time, postoperative pain and the need for additional hemostatic measures. In the literature, the risk of changes in ovarian reserve is also investigated, however it proved not significant and this was only a theoretical risk in the context of temporary clipping the infundibulopelvic artery, which is the main blood supply of the ovary. In this study, which will involve temporary clipping the utero-ovarian ligmant, there is no risk for a decrease in ovarian reserve.

ELIGIBILITY:
Inclusion Criteria:

Participants eligible for inclusion in this Trial must meet all of the following criteria:

1. Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures
2. Use of highly effective methods of birth control; defined as those that, alone or in combination, result in low failure rate (i.e., less than 1% per year) when used consistently and correctly; such as implants, injectables, combined oral contraceptives, some IUDs, true sexual abstinence (i.e. refraining from heterosexual intercourse during the entire period of risk associated with the Trial treatment(s)) or commitment to a vasectomised partner.
3. Female
4. Age: 18-50 years
5. Myomas, eligible for myomectomy, with the exclusion of FIGO 7-8 myomas.

Exclusion Criteria:

Participants eligible for this Trial must not meet any of the following criteria:

1. Any disorder, which in the Investigator's opinion might jeopardise the participant's safety or compliance with the protocol
2. Any prior or concomitant treatment(s) that might jeopardise the participant's safety or that would compromise the integrity of the Trial
3. Participation in an interventional Trial with an investigational medicinal product (IMP) or device
4. Patient refusal to participate in the Trial
5. (Possible) malignancy
6. any contra indication for a laparoscopic or robotic surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Peri-operative blood loss: Estimated blood loss | 1 week
  Multiple primary endpoints will be used to asses the blood loss:
  - Estimated blood loss >500 mL
Peri-operative blood loss: Hemoglobin drop perioperatively >2g/dL | 1 day
  Multiple primary endpoints will be used to asses the blood loss:
  - Hemoglobin drop perioperatively >2g/dL (difference between hemoglobin preoperatively and postoperatively)
Peri-operative blood loss: Need for peri-operative blood transfusion | 1 week
  Multiple primary endpoints will be used to asses the blood loss:
  - Need for peri-operative blood transfusion

SECONDARY OUTCOMES:
Hospitalisation time | 6 weeks
  Number of postoperative nights the patient had to stay in the hospital.
Operation time in minutes | 1 day
  Total surgical time, from the completion of anesthesia induction untill the end of surgery (in minutes)
Number of patients with complications postoperatively, graded by Clavien Dindo classification | 6 weeks
  The Clavien Dindo classification is a validated tool to quantitatively assess postoperative complications.
  Grade 0: No complications Grade 1: Any deviation from normal postoperative course, without requiring intervention Grade 2: Requiring pharmacological treatment Grade 3: Requiring surgical, endoscopic or radiological intervention Grade 4: Life-treathening complication requiring intermediate or intensive care Grade 5: Death of a patient
Number of patients requiring secondary hemostatic measures | 1 day
  Was there a need for non-routine hemostatic measures, such as:
  * Tranexamic acid
  * Misoprostol
  * Oxytocin
  * Embolisation
  * Local application of sealant patch or glue (e.g TachoSil or Tisseel)
  * Hysterectomy

CONTACTS AND LOCATIONS:
Overall Officials: Wouter Froyman, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (4):
- University Hospitals Leuven, Leuven, Belgium
- France (2):
  - Department of Gynecology and Obstetrics, Hopital Bichat, Paris
  - Service de gynécologie, Centre Hospitalier Universitaire de Rennes, Rennes
- Amsterdam UMC, locatie VUmc, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Williams VS, Jones G, Mauskopf J, Spalding J, DuChane J. Uterine fibroids: a review of health-related quality of life assessment. J Womens Health (Larchmt). 2006 Sep;15(7):818-29. doi: 10.1089/jwh.2006.15.818. PMID 16999637
- [Background] Pritts, E. A., & Olive, D. L. (2012). When Should Uterine Fibroids Be Treated? Current Obstetrics and Gynecology Reports. https://doi.org/10.1007/s13669-012-0010-y
- [Background] Stewart EA, Cookson CL, Gandolfo RA, Schulze-Rath R. Epidemiology of uterine fibroids: a systematic review. BJOG. 2017 Sep;124(10):1501-1512. doi: 10.1111/1471-0528.14640. Epub 2017 May 13. PMID 28296146
- [Background] Aendekerk, S., Verguts, J., Housmans, S., & Timmerman, D. (2019). Implementing robotic assisted myomectomy in surgical practice - a retrospective cohort study. Gynecological Surgery. https://doi.org/10.1186/s10397-019-1059-7
- [Background] Herrinton LJ, Raine-Bennett T, Liu L, Alexeeff SE, Ramos W, Suh-Burgmann B. Outcomes of Robotic Hysterectomy for Treatment of Benign Conditions: Influence of Patient Complexity. Perm J. 2020;24:19.035. doi: 10.7812/TPP/19.035. Epub 2019 Dec 18. PMID 31905335
- [Background] Winter ML, Leu SY, Lagrew DC Jr, Bustillo G. Cost comparison of robotic-assisted laparoscopic hysterectomy versus standard laparoscopic hysterectomy. J Robot Surg. 2015 Dec;9(4):269-75. doi: 10.1007/s11701-015-0526-z. Epub 2015 Jul 30. PMID 26530837
- [Background] Kongnyuy EJ, Wiysonge CS. Interventions to reduce haemorrhage during myomectomy for fibroids. Cochrane Database Syst Rev. 2014 Aug 15;2014(8):CD005355. doi: 10.1002/14651858.CD005355.pub5. PMID 25125317
- [Background] Ji L, Jin L, Hu M. Laparoscopic Myomectomy with Temporary Bilateral Uterine Artery Occlusion Compared with Traditional Surgery for Uterine Myomas: Blood Loss and Recurrence. J Minim Invasive Gynecol. 2018 Mar-Apr;25(3):434-439. doi: 10.1016/j.jmig.2017.06.032. Epub 2017 Sep 21. PMID 28943191
- [Background] Vercellino G, Erdemoglu E, Joe A, Hopfenmueller W, Holthaus B, Kohler C, Schneider A, Hasenbein K, Chiantera V. Laparoscopic temporary clipping of uterine artery during laparoscopic myomectomy. Arch Gynecol Obstet. 2012 Nov;286(5):1181-6. doi: 10.1007/s00404-012-2419-y. Epub 2012 Jun 20. PMID 22714065
- [Background] Hiratsuka D, Isono W, Tsuchiya A, Okamura A, Fujimoto A, Nishii O. The effect of temporary uterine artery ligation on laparoscopic myomectomy to reduce intraoperative blood loss: A retrospective case-control study. Eur J Obstet Gynecol Reprod Biol X. 2022 Aug 8;15:100162. doi: 10.1016/j.eurox.2022.100162. eCollection 2022 Aug. PMID 36035234
- [Background] Kim HC, Song T. Temporary simultaneous two-arterial occlusion for reducing operative blood loss during laparoscopic myomectomy: a randomized controlled trial. Surg Endosc. 2019 Jul;33(7):2114-2120. doi: 10.1007/s00464-018-6482-8. Epub 2018 Oct 17. PMID 30334154
- [Background] Coll S, Feliu S, Montero C, Pellise-Tintore M, Tresserra F, Rodriguez I, Barri-Soldevila PN. Evolution of laparoscopic myomectomy and description of two hemostatic techniques in a large teaching gynecological center. Eur J Obstet Gynecol Reprod Biol. 2021 Oct;265:181-189. doi: 10.1016/j.ejogrb.2021.08.023. Epub 2021 Aug 26. PMID 34509877
- [Background] Rothermel LD, Lipman JM. Estimation of blood loss is inaccurate and unreliable. Surgery. 2016 Oct;160(4):946-953. doi: 10.1016/j.surg.2016.06.006. Epub 2016 Aug 17. PMID 27544540
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912